CLINICAL TRIAL: NCT03514797
Title: Effect of a Single Prior Session of In-office Dental Bleaching on Time Required to Obtain Satisfactory Tooth Color With At-home Bleaching
Brief Title: Combined Dental Bleaching Protocols and Time Required to Achieve Satisfactory Color
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: André Luis Faria e Silva (Other)
Responsible Party: Sponsor-Investigator, André Luis Faria e Silva, Principal Investigator, Universidade Federal de Sergipe
Organization: Universidade Federal de Sergipe (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Combined bleaching
Record Dates: First submitted 2018-04-13; First posted 2018-05-02 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Tooth Discoloration
Keywords: Tooth bleaching; Hydrogen peroxide; Carbamide peroxide; Tooth Bleaching Agents
MeSH Terms: conditions — Tooth Discoloration | interventions — Bleaching Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined technique (Experimental): A single session of in-office tooth bleaching will be performed with 35% hydrogen peroxide for 45 minutes. Following, the teeth will be further bleached with customized trays filled with 10% carbamide peroxide and used for 1h per day.
  Interventions: Drug: Bleaching Agents
- At-home bleaching (Active Comparator): The teeth will be bleached only with customized trays filled with 10% carbamide peroxide and used for 1h per day.
  Interventions: Drug: Bleaching Agents

INTERVENTIONS:
Drug: Bleaching Agents — In-office tooth bleaching with 35% hydrogen peroxide in a single application of 45 minutes.
  Arms: Combined technique
Drug: Bleaching Agents — At-home tooth bleaching with 10% carbamide peroxide for 1 hour per day.

SUMMARY:
This parallel, randomized, and controlled clinical trial will assess the effect of a single prior session of in-office dental bleaching on time required to achieve satisfactory tooth color with at-home bleaching. Participants enrolled will randomly allocated to receive or not a single session of dental bleaching with 35% hydrogen peroxide applied for 45 min. Following, all participants will use customized trays filled with 10% carbamide peroxide for 1h per day until obtain satisfactory results. The primary outcome will be the number of days necessary to obtain satisfactory tooth color. Furthermore, tooth sensitivity and color changes measured with spectrophotometer will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Good general and oral health;
* Upper canines darker than the tab 2.5M2 at VITA Bleachedguide 3D-MASTER® (Vita-Zahnfabrik, Bad Sackingen, Germany) scale.

Exclusion Criteria:

* Presence of non-treated caries or periodontal disease;
* Prior tooth hypersensitivity;
* Presence of gingival recession;
* Teeth with cracked enamel or any hypoplasia;
* Patients using oral removable or fixed orthodontic appliances;
* Patients were pregnant or breastfeeding.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Time to tooth color satisfaction | up to 1 month after beginning the tooth bleaching procedures
  Time in days performing at-home bleaching necessary to participant reports that is satisfied with the tooth color obtained

SECONDARY OUTCOMES:
Color change | up to 1 month after beginning the tooth bleaching procedures
  Values of delta E measured with a spectrophotometer from color at baseline
Tooth sensitivity | 1, 2, 3, and 4 week after beginning the tooth bleaching procedures
  Maximum level of tooth sensitivity reported by participants using an analogue visual scale. The distance between the patient's marking and the no pain border was recorded in cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sergipe, Aracaju, Sergipe, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rezende M, Ferri L, Kossatz S, Loguercio AD, Reis A. Combined Bleaching Technique Using Low and High Hydrogen Peroxide In-Office Bleaching Gel. Oper Dent. 2016 Jul-Aug;41(4):388-96. doi: 10.2341/15-266-C. Epub 2016 Feb 26. PMID 26919081
- [Background] Cardoso PC, Reis A, Loguercio A, Vieira LC, Baratieri LN. Clinical effectiveness and tooth sensitivity associated with different bleaching times for a 10 percent carbamide peroxide gel. J Am Dent Assoc. 2010 Oct;141(10):1213-20. doi: 10.14219/jada.archive.2010.0048. PMID 20884923